CLINICAL TRIAL: NCT06622590
Title: A Single-center, Randomized, Blinded, and Positive Controlled Phase Ⅰ Clinical Trial of the Safety and Preliminary Immunogenicity of Quadrivalent Influenza Vaccine (split Virion) in People Aged 3 Years and Above
Brief Title: Phase I Clinical Trial of Quadrivalent Influenza Virus Split Vaccine
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Medical Biology, Chinese Academy of Medical Sciences (Other)
Collaborators: Guangxi Zhuang Autonomous Region Center for Disease Prevention and Control (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: 20221201_1
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Influenza, Human; Influenza a; Influenza Type B; Influenza Viral Infections
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: Three stages will be conducted according to the age-escalating principle.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (9):
- Intervention (Adults aged 18-59 years, one-dose) (Experimental): QIV in adults aged 18-59 years on Day 0
  Interventions: Biological: QIV
- Control (Adults aged 18-59 years, one-dose) (Active Comparator): Control vaccine in adults aged 18-59 years on Day 0
  Interventions: Biological: QIV control
- Intervention (Elders aged 60 years and above, one-dose) (Experimental): QIV in elders aged 60 years and above on Day 0
  Interventions: Biological: QIV
- Control (Elders aged 60 years and above, one-dose) (Active Comparator): Control vaccine in elders aged 60 years and above on Day 0
  Interventions: Biological: QIV control
- Intervention (Adolescents aged 9-17 years, one-dose) (Experimental): QIV in adolescents aged 9-17 years on Day 0
  Interventions: Biological: QIV
- Control (Adolescents aged 9-17 years, one-dose) (Active Comparator): Control vaccine in adolescents aged 9-17 years on Day 0
  Interventions: Biological: QIV control
- Intervention (Children aged 3-8 years, two-dose) (Experimental): QIV in children aged 3-8 years on Day 0 and Day 28
  Interventions: Biological: QIV
- Intervention (Children aged 3-8 years, one-dose) (Experimental): QIV in children aged 3-8 years on Day 0
  Interventions: Biological: QIV
- Control (Children aged 3-8 years, one-dose) (Active Comparator): Control vaccine n children aged 3-8 years on Day 0
  Interventions: Biological: QIV control

INTERVENTIONS:
Biological: QIV — Quadrivalent Influenza Virus Split Vaccine containing H1N1, H3N2, Bv, By antigens of 0.5ml for each dose
  Arms: Intervention (Adolescents aged 9-17 years, one-dose); Intervention (Adults aged 18-59 years, one-dose); Intervention (Children aged 3-8 years, one-dose); Intervention (Children aged 3-8 years, two-dose); Intervention (Elders aged 60 years and above, one-dose)
Biological: QIV control — Quadrivalent Influenza Virus Split Vaccine containing each type of antigens of 0.5ml for each dose
  Arms: Control (Adolescents aged 9-17 years, one-dose); Control (Adults aged 18-59 years, one-dose); Control (Children aged 3-8 years, one-dose); Control (Elders aged 60 years and above, one-dose)

SUMMARY:
This is a randomized, blinded, active-controlled phase I clinical trial to evaluate the safety and preliminary immunogenicity of the Quadrivalent Influenza Virus Split Vaccine (QIV) in subjects (aged 3 years and above). Primary endpoints are the occurrence of safety events after vaccination including the incidence of adverse events/adverse reactions within 30 minutes/7 days/30 days after immunization, as well as the incidence of serious adverse events/adverse relations within 6 months which will be defined as the secondary safety endpoint. Besides, the secondary immunogenicity endpoints are the geometric mean titers, geometric mean fold increases, seropositive rates, and seroconversion rates of anti-influenza virus HI antibodies for all types 30 days after immunization.

DETAILED DESCRIPTION:
This is a randomized, blinded, active-controlled phase I clinical trial to evaluate the safety and preliminary immunogenicity in 180 subjects (aged 3 years and above). Then 40 adults (aged 18-59 years), 40 elders (aged 60 years and above), 40 adolescents (aged 9-17 years), and 60 children (aged 3-8 years) are eligible for enrollment after assessing through the medical history and physical examination according to the principle of age escalating from adults to children.

40 adults in the first stage of the study will be randomly assigned to the vaccine and control cohort in a ratio of 1:1, that is, 20 subjects in such group will be injected with the experimental or active-controlled vaccine. The principal investigator and sponsors will conduct the safety evaluation by assessing the preliminary safety data within 7 days after the injection. If the results meet the criterion, the study will continue to the second stage after putting the record to IRB.

40 elders and 40 adolescents in the second stage of the study will be randomly assigned to the vaccine and control cohort in a ratio of 1:1, respectively, that is 40 subjects in such group will be injected with the experimental or active-controlled vaccine. The principal investigator and sponsors will conduct the safety evaluation by assessing the preliminary safety data within 7 days after the injection. If the results meet the criterion, the study will continue to the third stage after putting the record to IRB.

60 children in the third stage of the study will be randomly assigned to the 2-dose vaccine, 1-dose vaccine, and control group in a ratio of 1:1:1, that is 20 subjects in the 2-dose vaccine cohort will receive 2 doses of experimental vaccines in a 0,28 program, and 20 subjects in the 1-dose vaccine or control cohort will receive 1 dose of experimental or active-controlled vaccine. The principal investigator and sponsors will conduct the safety evaluation by assessing the preliminary safety data within 7 days after the injection. If the results meet the criterion, the study will continue to complete the second administration in the 2-dose vaccine cohort after putting the record to IRB.

The duration of intervention is no more than 1 month. With the 6-month safety monitoring after administration, the duration of the study is no more than 7 months.

For safety assessment, the observation and evaluation of adverse events from Day 0 to Day 30 after each dose will be conducted by diary/contact cards and investigators' phone calls. Besides, the observation and evaluation of serious adverse events up to 6 months after vaccination will be conducted by active reports by subjects' legal guardians, or investigators' phone calls as well as face-to-face visits. Meanwhile, subjects will be observed at the site for at least 30 minutes after each dose.

For laboratory examination, blood biochemistry, blood routine, and urine routine tests or urine pregnancy tests (if applicable) will be performed on Day 0 before vaccination as well as Day 4 after administration for all subjects.

For immunogenicity assessment, antibodies against all vaccine-related types of Influenza virus will be assessed in all subjects before vaccination and 30 days after full vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Age Requirement: volunteers aged 3 years and above at the time of enrollment
* Provision of Legal Identification: Volunteers and their legal guardians or appointed representatives must provide valid legal identification documents
* Informed Consent: Volutters, legal guardians, or appointed representatives of volunteers must have the capacity to understand the informed consent document and the research process, voluntarily participate, sign the informed consent form, and be able to comply with the requirements in the study as well as complete relevant visits on time.
* Temperature Requirement: Axillary body temperature is less than 37.3°C.
* Requirements for contraception: agree to take contraception actions in 6 months
* Previous Vaccination Requirements: (a) Received at least 1 dose of influenza vaccine within 1 year before screening in children aged 3-8 years; (b) Never received any influenza vaccine 1 year before screening in children aged 3-8 years.

Exclusion Criteria:

Subjects meeting any of the following exclusion criteria will be not eligible for enrollment.

* Subjects with a history of severe allergy to egg or egg protein, such as those who have had symptoms such as angioedema, dyspnea, chest distress, or repeated vomiting due to eating eggs, and even those who have used epinephrine or other emergency medical treatment, especially those who have symptoms immediately or within a short period (minutes to hours).
* Subjects with influenza illness (clinically, serologically, or microbiologically confirmed) within 6 months before screening and enrollment.
* Have received an influenza vaccine within 1 year before enrollment or scheduled to receive another influenza vaccine during the study period.
* Allergic to any component contained in the investigational vaccine, or previous history of severe allergic to any vaccine or drug, such as anaphylactic shock, laryngeal edema, anaphylactic purpura, thrombocytopenic purpura, local allergic necrosis reaction, dyspnea, angioedema, systemic rash and/or urticaria, etc.
* History of taking administration of a non-SARS-CoV-2 inactivated vaccine or subunit vaccine within 7 days before enrollment, or any live attenuated vaccine or SARS-CoV-2 vaccine within 14 days before enrollment, or subjects have scheduled to receive another vaccine within 1 month after receipt of the investigational vaccine
* Subjects with convulsion, epilepsy, encephalopathy (such as moderate to severe hypoxic-ischemic encephalopathy, intracranial hemorrhage, cerebral palsy, intracranial tumor, cerebral infarction, stroke, intracranial infection, etc.), psychiatric history or family history
* Have been diagnosed with a serious medical condition or congenital malformation that may interfere with the conduct or completion of the study (including but not limited to suffering from respiratory diseases such as asthma or during episodes of chronic bronchitis, Down syndrome, thalassemia, heart disease, severe cardiac arrhythmias, kidney disease, diabetes (diabetics with poor glycemic control or severe complications), autoimmune diseases, genetic allergies, Guillain-Barre syndrome, Crohn disease, malignancies, severe infectious/allergic skin diseases, etc.)
* Adults aged 18 years or older with medically uncontrolled abnormal blood pressure (systolic blood pressure ≥140mmHg and/or diastolic blood pressure ≥90mmHg or systolic blood pressure ≤ 90mmHg and/or diastolic blood pressure ≤ 60 mmHg)
* Subjects are acutely ill or in the acute phase of a chronic illness within 3 days before vaccination
* Subjects with fever (axillary temperature ≥37.3 ° C) within 3 days before vaccination or use of antipyretic, analgesic, or antiallergic medications
* Subjects with a hereditary bleeding tendency or coagulopathy, or a history of bleeding disorders
* Have received a blood transfusion or use of blood products within 6 months before enrollment, or planned to do so within 1 month after full immunization
* History of surgical removal of the spleen or other vital organs for any reason
* Use of any investigational or unregistered product (drug, vaccine, biological product, or device) other than a study vaccine within 3 months before enrollment or planned for use during the study
* Have treatment with immunosuppressive agents within 6 months before enrollment, such as long-term systemic glucocorticoid therapy (e.g., prednisone or a similar drug for more than 2 consecutive weeks within 6 months), but topical use (e.g., ointments, eye drops, inhalers, or nasal sprays) was allowed. Topical use should not exceed the recommended dose on the label or have any signs of systemic exposure
* Have been diagnosed with an infectious disease that may interfere with the conduct or completion of the study, such as active tuberculosis, hepatitis B, hepatitis C, human immunodeficiency virus (HIV) infection, etc
* Being lactating, pregnant (including a positive urine pregnancy test), or planning to become pregnant within 6 months of vaccination
* Subjects plan to move out of the local area before the end of the study or leave the local area for an extended period during the scheduled study visit
* Subjects with abnormal vital signs with clinical significance
* Investigators' Discretion: The final exclusion criterion is the discretion of investigators to determine whether a subject is suitable for participation in the study.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-10-13 (Actual); Primary Completion 2025-01-09 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Safety index - incidence of adverse events/adverse reactions | 0-30 minutes after the first dose vaccination
  Incidence of adverse events/adverse reactions after the first dose vaccination
Safety index - incidence of adverse events/adverse reactions | 0-30 minutes after the second dose vaccination
  Incidence of adverse events/adverse reactions after the second dose vaccination (applicable for the two-dose children cohort)
Safety index - incidence of adverse events/adverse reactions | Day 0 to 7 after the first dose vaccination
  Incidence of adverse events/adverse reactions after the first dose vaccination
Safety index - incidence of adverse events/adverse reactions | Day 0 to 7 after the second dose vaccination
  Incidence of adverse events/adverse reactions after the second dose vaccination (applicable for the two-dose children cohort)
Safety index - incidence of adverse events/adverse reactions | Day 0 to 30 after the first dose vaccination
  Incidence of adverse events/adverse reactions after the first dose vaccination
Safety index - incidence of adverse events/adverse reactions | Day 0 to 30 after the second dose vaccination
  Incidence of adverse events/adverse reactions after the second dose vaccination (applicable for the two-dose children cohort)

SECONDARY OUTCOMES:
Safety index - incidence of serious adverse events/adverse reactions | From the beginning of the vaccination up to 6 months after the last vaccination completed
  Incidence of serious adverse events/adverse reactions after vaccination
Immunogenicity index - seroconversion rates of HI antibody against all types | Between baseline and Day 30 after full vaccination
  Antibody assay will be performed using the hemagglutination inhibition test. Seroconversion will be defined as a change from seronegative (Antibody titers<1:40) to seropositive (Antibody titers≥1:40), or a ≥4-fold increase from baseline.
Immunogenicity index - Seropositive rates of HI antibody against all types | Day 30 after full vaccination
  Antibody assay will be performed using the hemagglutination inhibition test. Seropositive is defined as antibody titers≥1:40
Immunogenicity index - geometric mean titer (GMT) of HI antibody against all types | Day 30 after full vaccination
  Antibody assay will be performed using the hemagglutination inhibition test.
Immunogenicity index - geometric mean fold increases (GMT) of HI antibody against all types | Between baseline and Day 30 after full vaccination
  Antibody assay will be performed using the hemagglutination inhibition test.

CONTACTS AND LOCATIONS:
Overall Officials: Teng Huang, Principal Investigator — Guangxi Center for Disease Control and Prevention
Locations (1):
- Binyang Center for Disease Control and Prevention, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: No